CLINICAL TRIAL: NCT01504256
Title: Explorative Trial to Investigate Catumaxomab (Anti-EpCAM x Anti-CD3) for Treatment of Peritoneal Carcinomatosis in Patients With Gastric Adenocarcinomas Prior to Gastrectomy
Brief Title: Catumaxomab for Treatment of Peritoneal Carcinomatosis in Patients With Gastric Adenocarcinomas
Acronym: CatuNeo
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AIO-Studien-gGmbH (Other)
Collaborators: Neovii Biotech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AIO-STO-0110; 2010-024111-13 (EudraCT Number)
Record Dates: First submitted 2012-01-03; First posted 2012-01-05 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Gastric Adenocarcinoma With Peritoneal Carcinomatosis; Siewert Type II Adenocarcinoma of Esophagogastric Junction With Peritoneal Carcinomatosis; Siewert Type III Adenocarcinoma of Esophagogastric Junction With Peritoneal Carcinomatosis
Keywords: Adenocarcinoma; Esophagogastric Junction; Peritoneal Carcinomatosis; Catumaxomab; AIO-STO-0110
MeSH Terms: conditions — Adenocarcinoma; Peritoneal Neoplasms | interventions — catumaxomab; Fluorouracil; Leucovorin; Oxaliplatin; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- catumaxomab (Experimental): this arm was stopped. the antibody previously used as a study drug is not available at this time. patients will be randomized only into the standard arm
  [Catumaxomab: 4 intraperitoneal infusions of catumaxomab at an escalating dose of 10µg (d0), 20µg (d3), 50µg (d7), and 150µg (d10) and 7 days after the last catumaxomab infusion FLOT; 6 cycles q2w: Fluorouracil 2600 mg/m² as 24h infusion (d1) , leucovorin 200mg/m² (d1), oxaliplatin 85 mg{m² (d1), docetaxel 50 mg/m² (d1))
  Interventions: Drug: catumaxomab, Fluorouracil, leucovorin, oxaliplatin, docetaxel
- standard therapy (Active Comparator): FLOT; 6 cycles q2w:
  Fluorouracil 2600 mg/m² as 24h infusion (d1) leucovorin 200mg/m² (d1) oxaliplatin 85 mg{m² (d1) docetaxel 50 mg/m² (d1)
  Interventions: Drug: Fluorouracil, leucovorin, oxaliplatin, docetaxel

INTERVENTIONS:
Drug: catumaxomab, Fluorouracil, leucovorin, oxaliplatin, docetaxel — Catumaxomab: 4 intraperitoneal infusions of catumaxomab at an escalating dose of 10µg (d0), 20µg (d3), 50µg (d7), and 150µg (d10)
  and 7 days after the last catumaxomab infusion
  FLOT; 6 cycles q2w: Fluorouracil 2600 mg/m² as 24h infusion (d1) , leucovorin 200mg/m² (d1), oxaliplatin 85 mg{m² (d1), docetaxel 50 mg/m² (d1)
  Other Names: Catumaxomab + FLOT
  Arms: catumaxomab
Drug: Fluorouracil, leucovorin, oxaliplatin, docetaxel — FLOT; 6 cycles q2w:
  Fluorouracil 2600 mg/m² as 24h infusion (d1) leucovorin 200mg/m² (d1) oxaliplatin 85 mg{m² (d1) docetaxel 50 mg/m² (d1)
  Other Names: FLOT
  Arms: standard therapy

SUMMARY:
The purpose of this study is to determine the efficacy of catumaxomab by determination of the rate of macroscopic complete remissions of peritoneal carcinomatosis after treatment with one cycle (four doses) of catumaxomab followed by six cycles of routine neoadjuvant chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of resectable gastric adenocarcinoma or adenocarcinoma of the esophagogastric junction (type II and type III according to Siewerts classification)
* Macroscopic peritoneal carcinomatosis (stage P1-4 according to Gilly et al., appendix 1)
* Patients potentially eligible for gastrectomy after primary systemic (and intraperitoneal) treatment
* Signed and dated informed consent before the start of specific protocol procedures
* Age > 18 years
* ECOG Performance Status of 0 or 1
* Life expectancy of at least 12 weeks
* Adequate bone marrow, liver and renal function as assessed by the following laboratory requirements to be conducted within 7 days prior to screening

  * Hemoglobin > 10.0 g/dl
  * Leukocyte count > 4.000/μl; absolute neutrophil count (ANC) > 2.000/μl
  * Platelet count > = 100.000/µl
  * Total bilirubin < 1,5 times the upper limit of normal
  * ALT and AST < 3 x upper limit of normal
  * Alkaline phosphatase < 5 x ULN
  * Serum creatinine < 1.5 x upper limit of normal and creatinine clearance > 60 ml/min
* The patient is willing and able to comply with the protocol for the duration of the study, including hospital visits for treatment and scheduled follow-up visits and examinations

Exclusion Criteria:

* Distant metastasis other than peritoneal seedings
* Prior diagnosis of any malignancy not cured by surgery alone less than 5 years before study entry
* Clinically significant cardiovascular disease (incl. myocardial infarction, unstable angina, symptomatic congestive heart failure, serious uncontrolled cardiac arrhythmia) = < 1 year before enrolment
* History of HIV infection or chronic hepatitis B or C
* Active, clinically serious infections (> grade 2 NCI-CTC version 3.0)
* Pre-existing neuropathy > grade 1 (NCI CTCAE), except for loss of tendon reflex
* Patients with seizure disorder requiring medication (such as steroids or antiepileptics)
* History of organ allograft
* Patients undergoing renal dialysis
* Known hypersensitivity to any of the drugs given in the study; known hypersensitivity to murine (rat and/or mouse) proteins
* Any condition that is unstable or could jeopardize the safety of the patient and their compliance in the study
* Excluded therapies and medications, previous and concomitant:

  * Prior anti-cancer chemotherapy or immunotherapy.
  * Investigational drug therapy outside of this trial during or within 4 weeks of study entry
  * Major surgery within 4 weeks of starting the study, and patients must have recovered from effects of major surgery
* Pregnant or breast-feeding patients, or planning to become pregnant within 6 months after the end of treatment. Women of childbearing potential must have a negative pregnancy test performed within 7 days of the start of treatment. Women enrolled in this trial must use adequate barrier birth control measures during the course of the trial and for 6 months after the end of treatment
* Substance abuse, medical, psychological or social conditions that may interfere with the patient's understanding of the informed consent procedure, participation in the study or evaluation of the study results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2011-10; Primary Completion 2017-03 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Rate of macroscopic complete remissions of peritoneal carcinomatosis | Assessment after 14 - 18 weeks after start of treatment
  Macroscopic complete response (mCR) rate of the peritoneal lesions, as resulting from the second diagnostic laparoscopy or laparotomy performed after chemotherapy.

SECONDARY OUTCOMES:
Surgical resection rate (R0, R1, R2) | Assessment after 14 - 18 weeks after start of treatment
  All tumor evaluation is performed according to RECIST
Overall survival (OS) | Assessment over minimum 16 months up to 3 years
  The duration of overall survival (OS) will be determined by measuring the time interval from randomization to the date of death or last observation (censored).
Disease-free survival (DFS) | Assessment over minimum 16 months up to 3 years
  Disease-free survival (DFS) will be defined as the time from surgery, resulting in a R0 finding and macroscopic complete remission of PC, to the time of disease progression or relapse (according to RECIST) or death, or to the date of last assessment without any such event (censored observation). Patients with evidence of disease at surgery are counted as having the event at time = 0.
Progression-free survival (PFS) | Assessment over minimum 16 months up to 3 years
  Progression-free survival (PFS) will be defined as the time from randomization to the time of disease progression or relapse (according to RECIST) or death, or to the date of last assessment without any such event (censored observation).
Frequency, relationship, and severity of AEs | Assessment over minimum 16 months up to 3 years
Immunoreaction against tumor in tissue samples | 14 - 18 weeks
  blood and tumor tissue from every patient assed at 2time points. the first Laparoscopy (before randomization)and the second Laparoscopy (after chemotherapy)
Detection of disseminated tumor cells via PCR | 14 - 18 weeks
  blood and tumor tissue from every patient assessed at 2time points. the first Laparoscopy (before randomization) and the second Laparoscopy (after chemotherapy)

CONTACTS AND LOCATIONS:
Overall Officials: Florian Lordick, Prof. Dr., Principal Investigator — Universitäres Krebszentrum Leipzig (UCCL), Universität Leipzig, Medizinische Fakultät
Locations (1):
- Prof. Dr. F. Lordick, Leipzig, Germany

REFERENCES:
- See also: AIO - Working Group for Medical Oncology from the German Cancer Society — http://www.aio-portal.de